CLINICAL TRIAL: NCT03700385
Title: The IMPULSE Study: A Safety and Feasibility Study of the IOWA Approach Endocardial Ablation System to Treat Atrial Fibrillation
Brief Title: IMPULSE: A Safety and Feasibility Study of the IOWA Approach Endocardial Ablation System to Treat Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS0188
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Results first posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Patients undergoing catheter ablation of paroxysmal atrial fibrillation and meeting all protocol inclusion/exclusion criteria will be treated with the IOWA Approach Endocardial Ablation System.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- IOWA Approach Endocardial Ablation (Experimental): Subjects who are treated with the IOWA Approach Endocardial Ablation System for paroxysmal atrial fibrillation.
  Interventions: Device: IOWA Approach Endocardial Ablation System

INTERVENTIONS:
Device: IOWA Approach Endocardial Ablation System — Endocardial ablation using the IOWA Approach Endocardial Ablation System

SUMMARY:
IMPULSE is a prospective, single-arm, multi-center, safety and feasibility study evaluating the IOWA Approach Endocardial Ablation System (FARAPULSE, Inc.) for the treatment of paroxysmal atrial fibrillation.

DETAILED DESCRIPTION:
Patients undergoing catheter ablation for paroxysmal atrial fibrillation will be screened for enrollment per protocol inclusion and exclusion criteria. Enrolled patients will then undergo ablation using the IOWA Approach Endocardial Ablation System (FARAPULSE, Inc.). Subjects will be followed at 7 days, 30 days, 3 months, 6 months and 12 months with a blanking period for recurrent atrial fibrillation or atrial tachycardia of 3 months following the PEF catheter ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with PAF who have had at least one AF episode documented within one (1) year prior to enrollment. Documentation may include ECG, transtelephonic monitor (TTM), Holter monitor (HM), or telemetry strip.
2. Patients who have failed at least one antiarrhythmic drug (AAD; class I or III, or AV nodal blocking agents such as beta blockers and calcium channel blockers) as shown by recurrent symptomatic AF, or intolerance to the AAD or AV nodal blocking agents.
3. Patients who are ≥ 18 and ≤ 70 years of age on the day of enrollment.
4. Antero-posterior left atrial diameter ≤ 5.5 cm as documented by transthoracic echocardiography (TTE) or computed tomography (CT) within 3 months prior to the procedure.
5. Subject has no contraindications to intraoperative transesophageal echocardiography;
6. Left ventricular ejection fraction ≥40% as documented by TTE within 12 months prior to the procedure.
7. Received a standard cardiac work up and is an appropriate candidate for an investigational procedure as determined by study investigators.
8. Subject is willing and capable of providing Informed Consent to undergo study procedures and participate in all examinations and follow-up visits and tests associated with this clinical study.

Exclusion Criteria:

1. Patients on amiodarone at any time during the past 3 months prior to enrollment.
2. AF secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause.
3. AF episodes lasting > 7 days.
4. Previous ablation for AF.
5. Patient has a prosthetic heart valve.
6. Patient has a left atrial appendage device
7. Prior history of pericarditis or pericarditis within 3 months based on the TTE examination.
8. Subject is a woman of child bearing age
9. Prior history of rheumatic fever.
10. Prior history of medical procedure involving instrumentation of the left atrium (previous ablation, Atrial septal defect ASD closure, left atrial appendage occlusion)
11. History of severe chronic gastrointestinal problems involving the esophagus, stomach and/or untreated acid reflux
12. History of abnormal bleeding and/or clotting disorder.
13. Active malignancy or history of treated cancer within 24 months of enrollment.
14. Clinically significant infection or sepsis.
15. History of stroke or TIA within prior 6 months
16. New York heart Association (NYHA) class IIIb or IV congestive heart failure and/or any heart failure hospitalization within 3 months prior to enrollment.
17. Body mass index > 35.
18. Estimate glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2 or has ever received dialysis.
19. History of untreated and serious hypotension, bradycardia or chronotropic incompetence.
20. Any of the following within 3 months of enrollment:

    * Major surgery except for the index procedure
    * Myocardial infarction
    * Unstable angina
    * Percutaneous coronary intervention (e.g., CABG or PTCA)
    * Sudden cardiac death event
    * Left atrial thrombus that has not resolved as shown by TEE or CT
    * Implant of pacemaker, ICD or CRT.
21. Solid organ or hematologic transplant, or currently being evaluated for an organ transplant
22. History of pulmonary hypertension with Pulmonary systolic artery pressure >50 mm Hg, severe Chronic Obstructive Pulmonary Disease or restrictive lung disease.
23. Patients with any other significant uncontrolled or unstable medical condition (such as uncontrolled brady-arrhythmias, ventricular arrhythmias, hyperthyroidism or significant coagulation disorder).
24. Life expectancy less than one year.
25. Clinically significant psychological condition that in the physician's opinion would prohibit the subject's ability to meet the protocol requirements.
26. History of blood clotting or bleeding abnormalities.
27. Contraindication to anticoagulation (i.e., heparin, dabigatran, Vitamin K Antagonists such as warfarin).
28. Enrolled in another cardiac clinical study that would interfere with this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petr Neuzil, MD, PhD, Principal Investigator — Nemocnice Na Homolce
Locations (2):
- Nemocnice Na Homolce, Prague, Czechia
- CHU Bordeaux, Pessac, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reddy VY, Neuzil P, Koruth JS, Petru J, Funosako M, Cochet H, Sediva L, Chovanec M, Dukkipati SR, Jais P. Pulsed Field Ablation for Pulmonary Vein Isolation in Atrial Fibrillation. J Am Coll Cardiol. 2019 Jul 23;74(3):315-326. doi: 10.1016/j.jacc.2019.04.021. Epub 2019 May 11. PMID 31085321

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 40 subjects consented and were treated.
Pre-assignment Details: A total of 40 patients were enrolled (signed informed consent) and 40 subjects were treated at two (2) sites in Europe.
Period: Overall Study
Arm/Group | IOWA Approach Endocardial Ablation
Started | 40
Completed | 39
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | IOWA Approach Endocardial Ablation
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.2 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Czechia | 30
  France | 10

OUTCOME MEASURES:

1. Primary Outcome: The Primary Safety Endpoint for This Study is the Incidence of Early-onset (Within 7 Days of the PEF Ablation Procedure) Primary Adverse Events (AEs).
Description: The primary safety endpoint for this study is the incidence of early-onset (within 7 days of the PEF ablation procedure) primary adverse events (AEs).
  * Death
  * Myocardial infarction (MI)
  * Pulmonary vein (PV) stenosis†
  * Diaphragmatic paralysis
  * Atrio-esophageal fistula†
  * Transient Ischemic Attack (TIA)
  * Stroke/Cerebrovascular accident (CVA) Thromboembolism
  * Pericarditis requiring intervention (major)
  * Cardiac Tamponade/Perforation
  * Pneumothorax
  * Vascular Access Complications
  * Pulmonary edema
  * Hospitalization (initial and prolonged)*
  * Heart block
    * Excludes hospitalization (initial & prolonged) solely due to arrhythmia (AF/Atrial Flutter/Atrial Tachycardia) recurrence or due to non-urgent cardioversion (pharmacological or electrical).
      * Pulmonary vein (PV) stenosis or atrio-esophageal fistula that occurs greater than one week (7 days) post-procedure shall be deemed a Primary AE.
Time Frame: 7 days
Measure: Number; unit: percentage of participants
Arm/Group | IOWA Approach Endocardial Ablation
Number analyzed (Participants) | 40
percentage of participants | 2.5

2. Primary Outcome: Feasibility: Number of Patients With Pulmonary Vein Isolation
Description: Percentage of subjects achieving pulmonary vein isolation using the IOWA Approach Endocardial Ablation System.
Time Frame: 1 Day (Acute)
Measure: Count of Participants; unit: Participants
Arm/Group | IOWA Approach Endocardial Ablation
Number analyzed (Participants) | 40
Participants | 40

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | IOWA Approach Endocardial Ablation
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 7/40
Other Adverse Events (participants affected / at risk) | 7/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IOWA Approach Endocardial Ablation (N=40)
Atrial Fibrillation (Cardiac disorders) | 2 (2)
Atrial Tachycardia (Cardiac disorders) | 2 (2)
Cardiac Tamponade (Cardiac disorders) | 1 (1)
Calculus Urinary (Renal and urinary disorders) | 1 (1)
Arteriovenous Fistula (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IOWA Approach Endocardial Ablation (N=40)
Atrial Fibrillation (Cardiac disorders) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/85/NCT03700385/Prot_SAP_001.pdf